CLINICAL TRIAL: NCT06996171
Title: Comparative Efficacy of Magnesium Supplement and Melatonin Congener in Young Adults With Primary Insomnia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CMH Kharian Medical College (Other Government)
Responsible Party: Principal Investigator, Mushayada Irshad, Doctor, CMH Kharian Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CKMC/IERB/AC-00224
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Primary Insomnia
Keywords: Primary Insomnia; Magnesium supplement; Melatonin congener
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — magnesium diglycinate; Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A will receive magnesium supplements for 4 weeks (Oral, Tablet, Dose 500mg/day at night)
  Interventions: Drug: Magnesium glycinate
- Group B (Active Comparator): Group B will receive melatonin congener for 4 weeks (Oral, Tablet, Dose 10mg/day at night)
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Magnesium glycinate — Tab Magnesium glycinate 500mg will be given to one group for treatment of primary insomnia
  Arms: Group A
Drug: Melatonin — Tab Melatonin 10mg will be given to the other group for treatment of primary insomnia
  Arms: Group B

SUMMARY:
Sleep is essential for our overall health and well-being, much like food and water. It plays a vital role in numerous bodily functions. Many studies have been conducted to determine the efficacy of melatonin congeners and Mg supplements in patients with insomnia separately. This study aims to compare the efficacy of melatonin and magnesium supplements in young adults with primary insomnia. Most insomnia studies focus on older adults or individuals with comorbidities. Targeting otherwise healthy young adults brings age-specific relevance and novel insight.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* Gender: Male and Females (Non-pregnant & Non lactating)
* Diagnosed cases of primary insomnia according to following criteria:

  * Difficulty falling asleep, staying asleep or nonrestorative sleep
  * This difficulty is present despite adequate opportunity & circumstance to sleep
  * This impairment in sleep is associated with daytime impairment or distress
  * This sleep difficulty occurs at least 3 times per week and has been a problem for at least 1 month

Exclusion Criteria:

* Insomnia due to a known underlying cause
* Any psychiatric illness
* Active use of sedative hypnotics

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | 4 weeks
  ISI is a 7-item questionnaire used to determine the severity of insomnia.

CONTACTS AND LOCATIONS:
Locations (1):
- CMH Kharian Medical College, Kharan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
It will be decided after participants' consent whether to share their IPD or not.